CLINICAL TRIAL: NCT01318031
Title: Phase 1 Single Dose Open Label Study To Investigate The Potential DDI Between PF-00299804 And Paroxetine In Healthy Subjects
Brief Title: Study To Investigate The Potential Drug Drug Interaction (DDI) Between PF-00299804 And Paroxetine In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A7471021
Record Dates: First submitted 2011-02-17; First posted 2011-03-18 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
Keywords: DDI; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DDI (Experimental)
  Interventions: Drug: Period 1; Drug: Period 2

INTERVENTIONS:
Drug: Period 1 — Subjects will receive a single 45 mg dose of PF-00299804 on Day 1 of Period 1.
Drug: Period 2 — Subjects will receive a single 30 mg tablet of paroxetine once daily for 3 days (Days 1 to 3). Then, subjects will be co-administered a 45 mg single dose of PF-00299804 plus a single dose of 30 mg paroxetine on Day 4. Single 30 mg doses of paroxetine will be administered once daily for 6 days (Days 5-10).

SUMMARY:
Study of a drug drug interaction between Paroxetine and PF-00299804.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects must be extensive CYP2D6 metabolizers as determined by genotyping.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, dermatologic or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of depression or other potential for increased suicidality with paroxetine.
* Family or personal medical history of prolonged QTc, congenital deafness or sudden death, or 12-lead ECG with QTc>450 msec.
* A positive urine drug screen, use of tobacco or nicotine-containing products, or regular alcohol consumption exceeding 14 drinks/ week for females or 21 drinks/week for men within prior 6 months.
* Pregnant or nursing females and females of childbearing potential including those with tubal ligation. Women of 45 to 55 years of age who are postmenopausal must have confirmatory FSH test results at screening.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf of PF-00299804 when given alone in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks
Plasma AUCt of PF-00299804 when given alone in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks
Plasma Cmax of PF-00299804 when given alone in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks
Plasma AUCinf of PF-00299804 when given in combination with paroxetine in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks
Plasma AUCt of PF-00299804 when given in combination with paroxetine in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks
Plasma Cmax of PF-00299804 when given in combination with paroxetine in healthy volunteers who are extensive CYP2D6 metabolizers | 8 weeks

SECONDARY OUTCOMES:
Plasma CL/F of PF-00299804 in EM without paroxetine. | 8 weeks
Plasma Tmax of PF-00299804 in EM without paroxetine. | 8 weeks
Plasma t1/2 of PF-00299804 in EM without paroxetine. | 8 weeks
Plasma MRT of PF-00299804 in EM without paroxetine. | 8 weeks
Plasma CL/F of PF-00299804 in EM with paroxetine. | 8 weeks
Plasma Tmax of PF-00299804 in EM with paroxetine. | 8 weeks
Plasma t1/2 of PF-00299804 in EM with paroxetine. | 8 weeks
Plasma MRT of PF-00299804 in EM with paroxetine. | 8 weeks
Plasma AUCinf of PF-05199265 in EMs when given alone (if levels permit). | 8 weeks
Plasma AUCt of PF-05199265 in EMs when given alone (if levels permit). | 8 weeks
Plasma Cmax of PF-05199265 in EMs when given alone (if levels permit). | 8 weeks
Plasma Tmax of PF-05199265 in EMs when given in combination with paroxetine (if levels permit). | 8 weeks
Plasma t1/2 of PF-05199265 in EMs when given in combination with paroxetine (if levels permit). | 8 weeks
Overall safety profile as characterized by laboratory abnormalities, observed physical examination, vital signs, ECGs, and adverse event monitoring. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471021&StudyName=Study%20To%20Investigate%20The%20Potential%20Drug%20Drug%20Interaction%20%28DDI%29%20Between%20PF-00299804%20And%20Paroxetine%20In%20Healthy%20Subjects